CLINICAL TRIAL: NCT03170999
Title: Generation and Cognitive Testing of Informative and Suitable Items for a COPD Exacerbation Recognition Tool (CERT) for Detection of Exacerbations of COPD in Chinese Patients
Brief Title: Accurate Recognition of Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 201098
Record Dates: First submitted 2017-05-02; First posted 2017-05-31 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Airway Obstruction
Keywords: China; Cognitive testing; COPD exacerbation; CERT
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subjects included in Focus groups: Approximately 45 subjects with COPD will participate in the focus group interviews for item identification. The group may contain subjects who are functionally illiterate and at least one third women will be recruited.
  Interventions: Other: Focus group interview
- Subjects included in cognitive interviews: Approximately 9 subjects with COPD will be involved in cognitive interviews and will be asked to respond to all of the items in the draft item set.
  Interventions: Other: Draft item set
- Subjects included in candidate item set: Approximately 150 subjects with COPD will respond to the questions in candidate item set.
  Interventions: Other: Candidate item set

INTERVENTIONS:
Other: Focus group interview — Focus group interviews will take place to discuss the key domains of COPD exacerbation which then will be used in the formation of the draft item set.
  Groups: Subjects included in Focus groups
Other: Draft item set — Items that form the draft item set will be subject to cognitive debriefing. Questions in the draft item set will collect information on whether the subjects with COPD have experienced that item during an exacerbation. Changes in this draft set will result in the formation of candidate item set.
  Groups: Subjects included in cognitive interviews
Other: Candidate item set — Item reduction will be done using candidate item set and the subjects will be asked to respond to the candidate items on a 4-point scale in terms of how that item changed with the onset of the last episode. Item reduction will take into account frequency and magnitude of items, floor and ceiling items and consistency between regions. The candidate item set will then be used for generation of CERT.
  Groups: Subjects included in candidate item set

SUMMARY:
It has been observed that COPD exacerbations are under-reported in China. One of the reasons for this is Chinese subjects with COPD cannot describe the symptoms of exacerbation mentioned in English. Hence this study aims to create a tool called CERT that will help Chinese physicians and subjects with COPD to recognize and report exacerbations. The study will be carried out in 4 stages: item identification, cognitive briefing, item reduction and creation of final CERTs. Two CERTs will be prepared, one for subjects with COPD and another for physicians. A total of approximately 200 subjects will be included in the study and each subject will contribute to only one step.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of age greater than or equal to 40 years.
* Spirometrically confirmed COPD according to diagnostic criteria in Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2016.
* A treated exacerbation of COPD within 3 months prior to the study visit.
* Willing and able to provide informed consent, and able to participate in focus groups or cognitive interviews.
* Literacy is not a requirement for any of the groups.

Exclusion Criteria:

* Current diagnosis of asthma or clinically relevant bronchiectasis. Note: Subjects with Asthma COPD Overlap Syndrome (ACOS) are eligible.
* Subjects with a concurrent significant, uncontrolled, active medical condition or disease state of other organ diseases or systematic diseases; psychiatric condition; cognitive impairment or any other reasons that in the investigator's opinion, would place subjects at risk or interfere with study evaluation or affect participation in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects having COPD attending the outpatient respiratory specialist clinics of tier 3 hospitals for their disease will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
COPD symptom item set to identify common phrases of COPD exacerbation | Day 1
  The most frequently used items to describe the symptomatic characteristics of the onset of an exacerbation will be identified from COPD symptom item set.
Preparation of COPD Exacerbation Recognition tool (CERT) | Day 1
  Two simple educational hand-outs called CERT will be prepared, one for the subjects with COPD and the other for the physicians which will help Chinese physicians and subjects in recognizing and reporting COPD exacerbations.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- China (3):
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Shenyang